CLINICAL TRIAL: NCT06461962
Title: Rural Community Peer Partnerships for Improving Methamphetamine-Associated Heart Failure Screening and Engagement
Acronym: PEER-Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Washington (Other); Bay Area First Step (Unknown)
Responsible Party: Principal Investigator, Brian L Chan, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00026150
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Methamphetamine Use; Heart Failure
Keywords: Screening; Implementation Science; Heart Failure; Addiction; Stimulants; Health Services; Community Engaged Research
MeSH Terms: conditions — Heart Failure; Behavior, Addictive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer-supported Treatment as Usual (Active Comparator): Participants will receive a peer-supported referral to a local primary care provider who will create a plan to treat the participants heart failure.
  Interventions: Other: Treatment as Usual
- Peer-Supported Telehealth Cardiology (Experimental): Participants will receive a virtual consultation with a cardiovascular specialist, referral for a locally performed echocardiogram (ECG), and transitional care management facilitated by a remote nurse care manager and the peer to treat the participants heart failure.
  Interventions: Other: Telehealth-Cardiology

INTERVENTIONS:
Other: Treatment as Usual — Peer-facilitated referral to a local primary care provider to follow-up their screening results.
  Arms: Peer-supported Treatment as Usual
Other: Telehealth-Cardiology — Peer-facilitated virtual consultation with cardiovascular specialist, for follow-up of their screening results. Activities may include: referral for a locally performed testing including echocardiogram and additional blood work, and transitional care management facilitated by a remote nurse care manager and the peer
  Referral for a locally performed testing including echocardiogram
  Transitional care management facilitated by a remote nurse care manager and the peer
  Arms: Peer-Supported Telehealth Cardiology

SUMMARY:
The goal of PEER-Heart is to implement and assess feasibility and preliminary effectiveness of a community peer-facilitated screening for methamphetamine-associated heart failure (MAHF) and linkage to evidence-based cardiology care for people who use methamphetamine in rural areas.

DETAILED DESCRIPTION:
Methamphetamine use has increased across the US in the midst of the opioid crisis, with rates of methamphetamine use in rural communities exceeding that in urban areas. Nationwide, methamphetamine-related hospitalizations increased 270% between 2007 and 2015, along with associated costs, lengths of stay and mortality. Methamphetamine-associated heart failure (MAHF) hospitalizations increased 12-fold over this time period; it is associated with worse symptoms (e.g. ejection fraction) and decreased adherence to guideline-directed medical therapy (GDMT) compared to heart failure not associated with methamphetamine use.

Despite the increased risk of heart failure and overdose for people who use methamphetamine in rural areas, interventions to improve engagement in cardiac screening and treatment services are underdeveloped. Multiple barriers decrease access to cardiac care in rural communities, including social determinants of health and health systems care delivery barriers. Stigma and distrust of healthcare providers, particularly in rural communities are known barriers to engaging in medical care-COVID-19 has only worsened this gap for people who use drugs.

Team-based cardiology care interventions can improve outcomes for people with heart failure, including one multi-disciplinary program that focused on methamphetamine-associated heart failure MAHF. However, these interventions have been tested in urban, higher resourced settings than those typical in rural communities. Interventions for screening and linkage to care for people who use drugs in rural areas with MAHF have not been developed.

The "experiential credentialing" afforded by peer recovery support specialists ("peers") offers a unique opportunity to reach, engage, and retain non-treatment-seeking people using drugs. The PEER-Heart study extends the role of peers as trusted community health workers in rural communities to improve MAHF screening and linkage to cardiology care. Increasing evidence reports feasibility, acceptability, and effectiveness of telehealth interventions in rural communities including cardiology services and retention in substance use treatment. Virtual visits for heart failure demonstrate promise in improving follow-up care though more study is warranted to demonstrate clinical outcomes effectiveness, and ensure these interventions do not worsen existing health inequities and the rural digital divide, particularly in minoritized groups.

The PEER-Heart study aims to demonstrate feasibility of screening of MAHF and linkage to evidence-based cardiology care for people who use methamphetamine in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Patient-defined regular use of methamphetamine in the last year
* Any methamphetamine use in the past 30 days
* Age 18 years or older
* No client-reported diagnosis of heart failure
* Able to communicate in English
* Screen positive for potential methamphetamine-associated heart failure (MAHF) defined as B type natriuretic peptide (BNP) ≥50 pg/ml, or QRS width ≥120ms, or presence of any clinical heart failure symptoms

Exclusion Criteria:

* Self-reported engagement in medical care for heart failure in past 6 months.
* Actively taking medications for heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Linkage to cardiology care | 2 months
  Proportion of participants who are engaged in cardiac care at 2 months after screening.

SECONDARY OUTCOMES:
Linkage to diagnostic echocardiogram | 2 months
  Proportion of participants who complete a diagnostic echocardiogram within 2 months after randomization.
Goal Directed Medical Therapy (GDMT) prescribed | 6 months
  Proportion of eligible patients who are on any GDMT at 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chan, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared following data lock with the data coordinating center at University of Washington.
Time Frame: Following data lock.